CLINICAL TRIAL: NCT05665777
Title: The Effectiveness and Safety of Qingyan Lihou Decoction for the Treatment of Chronic Pharyngolaryngitis: A Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Chinese Medicine for Treating Chronic Pharyngolaryngitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Lin Zhixiu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP study
Record Dates: First submitted 2022-12-18; First posted 2022-12-27 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Chronic Pharyngolaryngitis (Disorder)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Qingyan Lihou Decoction) (Experimental): It consists of 22 kinds of Chinese medicine as ingredients. It was prepared in granule form.
  Interventions: Drug: Qingyan Lihou Decoction
- Placebo (Placebo Comparator): The placebo medication is composed of starch and an edible pigment and will be matched as closely as possible to the appearance and taste of Qingyan Lihou Decoction granules.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Qingyan Lihou Decoction — Chinese medicine granules
  Other Names: Active treatment
  Arms: Active treatment (Qingyan Lihou Decoction)
Other: Placebo — Placebo granules
  Arms: Placebo

SUMMARY:
A randomized, double-blinded, placebo-controlled clinical trial using a Chinese Medicine formula in treating Chronic pharyngolaryngitis. Subjects will be randomized into a treatment group or placebo group for 8 weeks, and then followed by an 8-week post-treatment visit.

DETAILED DESCRIPTION:
Chronic pharyngolaryngitis (CP), also known as chronic pharyngitis, is defined as the inflammation of the pharynx, which is at the back of the throat. CP is a common disease characterized by dry throat, sore throat, pharyngeal itching, dry cough, and difficulty in swallowing. In Western medicine, common treatment regimens for CP include lozenges, antibiotics, lasers, and cryotherapy. However, the above treatment modalities may not be effective, and the disease is likely to bounce back repeatedly.

Chinese medicine has been used for the treatment of CP for a long time. Many studies have shown that treatment using Chinese herbal medicine is effective in relieving the symptoms of CP.

This study is to evaluate the efficacy and safety of oral Qingyan Lihou Decoction in relieving the clinical symptoms of patients with CP.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or above (Chinese subjects only);
* Persistent symptoms of pharyngitis (sore throat, globus, dry throat, dry cough, throat irritation) for more than 3 weeks;
* Determined to be the following Chinese medicine syndromes by Registered Chinese Medicine Practitioners (RCMPs): Wind-heat invading the upper-jiao, or phlegm heat or Yin deficiency;
* Visual analog scale (VAS) score for pain ≥ 50 mm;
* Numeric rating scale (NRS) ≥ 6; and
* Be able to give voluntary written informed consent.

Exclusion Criteria:

* Known severe medical conditions, such as cardiovascular, liver or renal dysfunction, diabetes mellitus, cancers, cerebrovascular diseases, blood system diseases;
* Concomitant use of steroids, nonsteroidal anti-inflammatory drugs (NSAIDs), anticoagulants, and immunotherapy within the past week;
* Impaired hematological profile and liver / renal function exceed the upper limit of the reference value by 2 times;
* Known Allergic rhinitis;
* Known Gastroesophageal Reflux Disease (GERD);
* Known cancer or suspected cancer of throat/oesophagus;
* Mechanical obstruction of the throat accountable for the symptoms;
* Known alcohol and/or drug abuse;
* Known allergic history to any Chinese herbal medicines; and
* Subjects who are known pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
The resolution rate of the clinical symptoms of CP | 8 weeks
  Measure the resolution rate of the clinical symptoms at week 8. According to the "Guiding Principles for Clinical Research of Chinese Medicines", the degree of clinical symptom is divided into 4 grades: asymptomatic, mild symptom, moderate symptom, and severe symptom, with a score of 0~3.
Improvement of laryngeal signs | 8 weeks
  Observe the improvement of laryngeal signs via Flexible nasopharyngolaryngoscopy examination

SECONDARY OUTCOMES:
Complete remission rate of Globus | 8 weeks
  The rate of remission of the main clinical symptom Globus at week 8. According to the "Guiding Principles for Clinical Research of Chinese Medicines" [16], the degree of clinical symptom is divided into 4 grades: asymptomatic, mild symptom, moderate symptom, and severe symptom, with a score of 0~3.
Complete remission rate of Globus symptom | 16 weeks
  The rate of remission of main clinical symptom Globus at week 16. According to the "Guiding Principles for Clinical Research of Chinese Medicines" [16], the degree of clinical symptom is divided into 4 grades: asymptomatic, mild symptom, moderate symptom, and severe symptom, with a score of 0~3.
Visual analogue scale (VAS) of Globus symptom | 8 weeks
  Difficulty in swallowing is assessed using a VAS, which is 100 mm in length (100-mm VAS) anchored by two verbal descriptors, one for each extreme symptom (0 mm = not difficult, 100 mm = very difficult)
Visual analogue scale (VAS) of Globus symptom | 16 weeks
  Difficulty in swallowing is assessed using a VAS, which is 100 mm in length (100-mm VAS) anchored by two verbal descriptors, one for each extreme symptom (0 mm = not difficult, 100 mm = very difficult)
Change of Numeric rating scale of sore throat | 8 weeks
  Intensity of sore throat will be assessed using an 11-point numeric rating scale (11-point NRS) with 0 representing one pain extreme (no pain) and 10 representing the other pain extreme (most severe pain)
Change of Numeric rating scale of sore throat | 16 weeks
  Intensity of sore throat will be assessed using an 11-point numeric rating scale (11-point NRS) with 0 representing one pain extreme (no pain) and 10 representing the other pain extreme (most severe pain)
Changes of serum level of cytokines | 8 weeks
  Blood samples will be taken to detect the serum level of C reactive protein (CRP), Erythrocyte Sedimentation Rate (ESR), Complete blood count (CBC), White blood cell (WBC), and Antinuclear antibody (ANA) using enzyme-linked immunosorbent assay (ELISA) kits. These are the markers for inflammatory response and severity. The higher the value, the more severity of the symptoms.
Changes of serum level of cytokines | 16 weeks
  Blood samples will be taken to detect the serum level of C reactive protein (CRP), Erythrocyte Sedimentation Rate (ESR), Complete blood count (CBC), White blood cell (WBC), and Antinuclear antibody (ANA) using enzyme-linked immunosorbent assay (ELISA) kits. These are the markers for inflammatory response and severity. The higher the value, the more severity of the symptoms.
Changes of laryngeal hypersensitivity questionnaire (LHQ) | 8 weeks
  LHQ contains 14 items with a 7-point Likert frequency response scale where 1 equates to all of the time and 7 equates to none of the time. 14 items will be divided into 3 categories, which is obstruction, pain and throat tickle. Average score of each category will be obtained and the total LHQ score will be the sum of those average scores.
Changes of laryngeal hypersensitivity questionnaire (LHQ) | 16 weeks
  LHQ contains 14 items with a 7-point Likert frequency response scale where 1 equates to all of the time and 7 equates to none of the time. 14 items will be divided into 3 categories, which is obstruction, pain and throat tickle. Average score of each category will be obtained and the total LHQ score will be the sum of those average scores.
Changes of oral microbiome | 8 weeks
  The saliva sample will be collected from subjects, and it will be examined according to the protocol of the Microbiome Saliva DNA Kit.
Changes of oral microbiome | 16 weeks
  The saliva sample will be collected from subjects, and it will be examined according to the protocol of the Microbiome Saliva DNA Kit.
Changes in Sore Throat Assessment Tool-10 (STAT-10) | 8 weeks
  The STAT-10 is the first validated tool for measuring the intensity and duration of symptoms from the perspective of sore throat patients and for quantifying and comparing different treatment modalities in acute pharyngotonsillitis (APT) patients. STAT-10 contains 10-item questionnaire using a five-point Likert scale. The higher the score, the more severity of the symptoms.
Changes in Sore Throat Assessment Tool-10 (STAT-10) | 16 weeks
  The STAT-10 is the first validated tool for measuring the intensity and duration of symptoms from the perspective of sore throat patients and for quantifying and comparing different treatment modalities in acute pharyngotonsillitis (APT) patients. STAT-10 contains 10-item questionnaire using a five-point Likert scale. The higher the score, the more severity of the symptoms.
Changes in Eating Assessment Tool-10 (EAT-10) | 8 weeks
  It consists of ten statements that a patient rates on a scale of 0-4, with 0=no problem to 4=severe problem. The score is 0 to 40. The higher the score, the more severity of the swallowing difficulty.
Changes in Eating Assessment Tool-10 (EAT-10) | 16 weeks
  It consists of ten statements that a patient rates on a scale of 0-4, with 0=no problem to 4=severe problem. The score is 0 to 40. The higher the score, the more severity of the swallowing difficulty.
Adverse event related to the study treatment | From baseline to week 16
  Any adverse event will be recorded during the study period, it will be graded by CTCAE.
Changes in 36-Item Short Form Survey Instrument (SF-36) | 8 weeks
  It will be used to assess the patient's health status using 8 different dimensions including vitality, physical functioning, bodily pain, general health perceptions, role limitations due to physical health, role limitations due to emotional health, social role functioning and mental health. The possible score ranges from 0 to 100 points whereby 0 points represent the greatest possible limitation of health, while 100 points represent the absence of health restrictions.
Changes in 36-Item Short Form Survey Instrument (SF-36) | 16 weeks
  It will be used to assess the patient's health status using 8 different dimensions including vitality, physical functioning, bodily pain, general health perceptions, role limitations due to physical health, role limitations due to emotional health, social role functioning and mental health. The possible score ranges from 0 to 100 points whereby 0 points represent the greatest possible limitation of health, while 100 points represent the absence of health restrictions.

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiu Lin, Principal Investigator — Hong Kong Institute of Integrative Medicine
Locations (1):
- Hong Kong Institute of Integrative Medicine, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No